CLINICAL TRIAL: NCT04186091
Title: Perfusion Index Predicts Post-spinal Hypotension in Obese Parturients for Cesarean Section-A Prospective Observational Study
Brief Title: Perfusion Index Predicts Post-spinal Hypotension in Obese Parturients for Cesarean Section
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Other Study IDs: N-5- 2017
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Perfusion Index Predicts Post-spinal Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: correlation between baseline perfusion index and decrease in systolic blood pressure post spinal induction — correlation between baseline perfusion index and decrease in systolic blood pressure post spinal induction

SUMMARY:
Hypotension is a common adverse effect of spinal anesthesia during caesarean section especially in obese patients.

The aim of this study is to find out the correlation between baseline PI and post spinal hypotension in obese parturient.

DETAILED DESCRIPTION:
Abstract Background Hypotension is a common adverse effect of spinal anesthesia during caesarean section especially in obese patients.

The aim of this study is to find out the correlation between baseline PI and post spinal hypotension in obese parturient.

Methods After approval of ethical committee and written informed consent, fifty Parturients aged between 18- 40 years, ASA I and II with term singleton pregnancies with BMI between 25 &40 admitted for cesarean section under spinal anesthesia were recruited in this prospective, observational study. The primary outcome is the correlation between baseline perfusion index and post spinal hypotension. The secondary outcome is the correlation between BMI and the incidence of hypotension after spinal anesthesia. Heart rate, blood pressure, perfusion index before and after spinal induction using Masimo device, level of sensory block, dose of ephedrine required to correct hypotension, dose of atropine required to correct bradycardia, incidence of nausea, vomiting and shivering were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Fifty parturient
* Aged between 18- 40,
* ASA I and II
* With term singleton pregnancies
* With 25 ≥ BMI≤ 40
* Conducted for cesarean section under spinal anesthesia

Exclusion Criteria:

* Emergency cases,
* Placenta previa,
* Preeclampsia,
* Cardiovascular and cerebrovascular diseases,
* Patient with contraindication for regional anesthesia
* Patient with peripheral vascular diseases as DVT.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: After approval of ethical committee and written informed consent, fifty Parturients aged between 18- 40 years, ASA I and II with term singleton pregnancies with BMI between 25 &40 admitted for cesarean section under spinal anesthesia were recruited in this prospective, observational study. The primary outcome is the correlation between baseline perfusion index and post spinal hypotension. The secondary outcome is the correlation between BMI and the incidence of hypotension after spinal anesthesia. Heart rate, blood pressure, perfusion index before and after spinal induction using Masimo device, level of sensory block, dose of ephedrine required to correct hypotension, dose of atropine required to correct bradycardia, incidence of nausea, vomiting and shivering were recorded.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
correlation between baseline perfusion index and post spinal decrease in systolic blood pressure | 24 hours Postoperative
  correlation between baseline perfusion index and post spinal decrease in systolic blood pressure

SECONDARY OUTCOMES:
correlation between BMI and the incidence of post-spinal hypotension | 24 hours Postoperative
  correlation between BMI and the incidence of post-spinal hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Study Director — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till submission